CLINICAL TRIAL: NCT02744053
Title: Multimodality Breast Imaging for the Assessment of Tumor Response to Neoadjuvant Chemotherapy in Triple Negative Breast Cancer Patients
Brief Title: DCE-MRI and MBI in Assessing Tumor Response to Chemotherapy in Patients With Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-0816; NCI-2016-00715 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0816 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-04-05; First posted 2016-04-20 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Progesterone Receptor Negative; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (DCE-MRI, MBI) (Experimental): Patients undergo DCE-MRI over 45-60 minutes. Patients receive technetium Tc-99m sestamibi via injection, and after 5 minutes patients undergo MBI scan over 1 hour. Both DCE-MRI and MBI are performed at the time of enrollment, at the end of anthracycline therapy, and at the conclusion of NAC before surgery. All patients also undergo standard of care imaging with DM and US (at the same time points if the treating doctor chooses to do so).
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Laboratory Biomarker Analysis; Radiation: Scintimammography; Drug: Technetium Tc-99m Sestamibi

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Scintimammography — Undergo MBI
  Other Names: Breast-Specific Gamma Imaging; MBI; Miraluma Scan; Miraluma Test; Molecular Breast Imaging; Nuclear Medicine Breast Imaging; sestamibi breast imaging; Sestamibi Scintimammography
Drug: Technetium Tc-99m Sestamibi — Given via injection
  Other Names: Cardiolite; Miraluma; Tc 99m Sestamibi; Tc-99m MIBI; Tc99m Sestamibi

SUMMARY:
This early phase I trial studies how well dynamic contrast enhanced molecular resonance imaging (DCE-MRI) and technetium-Tc99m sestamibi molecular breast imaging (MBI) work in assessing tumor response to chemotherapy in patients with triple negative breast cancer (TNBC) who are undergoing chemotherapy. Investigational imaging scans such as MBI and DCE-MRI may help researchers predict which patients may respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the predictive value of advanced imaging modalities Tc99m sestamibi (technetium Tc-99m sestamibi) molecular breast imaging (MBI) and dynamic contrast enhanced (DCE) magnetic resonance imaging (MRI) for neoadjuvant chemotherapy (NAC) response in triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To evaluate and compare the ability all imaging modalities including standard of care digital mammogram (DM) and ultrasound (US) as well as novel modalities DCE-MRI and MBI to assess and predict response to neoadjuvant chemotherapy (NAC) in patients with triple negative breast cancer (TNBC).

EXPLORATORY OBJECTIVES:

I. To determine effect of molecular subtype of TNBC on diagnostic performance of different types of imaging modalities in predicting treatment response.

II. To determine the Utility of Dynamic Tc99m sestamibi MBI and DCE-MRI together with molecular profiling to identify a subgroup of chemoresistant TNBC patients.

OUTLINE:

Patients undergo DCE-MRI over 45-60 minutes. Patients receive technetium Tc-99m sestamibi via injection, and after 5 minutes patients undergo MBI scan over 1 hour. Both DCE-MRI and MBI are performed at the time of enrollment, at the end of anthracycline therapy, and at the conclusion of NAC before surgery. All patients also undergo standard of care imaging with DM and US (at the same time points if the treating doctor chooses to do so).

ELIGIBILITY:
Inclusion Criteria:

* The patient has proven TNBC, defined by standard pathologic assays as negative for estrogen receptor (ER) and progesterone receptor (PR) (< 10% tumor staining) and negative for human epidermal growth factor 2 (HER2) (immunohistochemistry [IHC] score < 3, gene copy number not amplified)
* TNBC patients who are previously untreated and enrolled in the prospective Institutional Review Board (IRB) approved clinical trial: 2014-0185
* Patients who are able to understand and give consent to participating in the study

Exclusion Criteria:

* Is pregnant (confirmed by the patient as imaging clinic standard of care) or nursing mother
* Has lesions involving chest wall
* Has known allergy to Tc99m sestamibi
* Has known contraindications to MRI
* Has contraindication to MRI contrast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in volume of index tumors and estimated area under receiver operating characteristic (ROC) curves assessed by digital mammogram, ultrasound, dynamic contrast enhanced molecular resonance imaging (DCE-MRI) and molecular breast imaging (MBI) | Up to 4 years
  The ability to assess and predict response will be compared among the imaging modalities and with standard pathological evaluation. These volume changes will be correlated with residual cancer burden (RCB) status after surgery and will be used to classify patients into predicted responder or non-responder categories. Predictive accuracies among the imaging modalities will be compared using paired ROC curve analyses.
Percent change in tumor volume assessed by dynamic Tc99m-sestamibi MBI | up to 6 months
  The index tumor will be measured on both cranial-caudal (CC) and medio-lateral oblique (MLO) views and 3 dimension will be recorded. The percentage change in volume at time points 2 and 3 relative to baseline imaging (time point 1) will be calculated. Data acquisition and image processing algorithms will be developed from having conjugate views of the breast in the MBI examination. Appropriate methods to correct the image from loss of contrast due to scatter and loss of signal from photon attenuation as it transits breast tissue will be explored and implemented. Will investigate the correlations of absolute and relative values of baseline standardized uptake value (SUVb) with pathological tumor response.
Tumor response assessed by pathological examination | Up to 4 years
  Correlations of pathological response with absolute and relative values of MBI SUVb will be investigated. The longest dimension of the residual tumor will be measured. If only foci of disease are seen the longest dimension of tumor cell distribution will be measured. The M D Anderson Cancer Center (MDACC) Residual Cancer Burden Calculator will be used to categorize cancer burden: RCB-0 (no residual disease in breast or in lymph nodes), RCB-1 (minimal residual disease), RCB-2 (moderate residual disease), or RCB-3 (extensive residual disease).

OTHER OUTCOMES:
Utility of molecular breast imaging (MBI) and dynamic contrast enhanced molecular resonance imaging (DCE-MRI) together with molecular profiling to identify a subgroup of chemoresistant triple negative breast cancer (TNBC) patients | up to 6 months
  Assessed by baseline SUVb and baseline genomic signature. Will fit one logistic regression model with baseline SUVb and baseline genomic signature as covariates and response to the upfront chemotherapy as the endpoint and one model with baseline DCE-MRI tumor volume and baseline genomic signature as covariates and response to the upfront chemotherapy as the endpoint. Will assess the predictive accuracy of this model by estimating the area under the ROC curve using the predicting response probability and the observed response outcome. ROC curves will be generated for each modality and each TNBC molecular subtype and compute the areas under these curves along with 95% confidence intervals. Will determine a cut-point in the predicted probabilities to classify patients as predicted responders and non-responders based an appropriate trade-off between sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Gaiane M Rauch, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org